CLINICAL TRIAL: NCT05542316
Title: Validation of the Polymyalgia Rheumatica Activity Score for Determination of Disease Activity
Brief Title: Validation of the PMR Activity Score and Evolution of Patient-reported Outcomes in Patients With Polymyalgia Rheumatica
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66638
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a final diagnosis of PMR

SUMMARY:
Polymyalgia rheumatica (PMR) is a systemic inflammatory disease that affects elderly people. It is characterized by pain and morning stiffness in the shoulders, pelvic girdles and neck. Glucocorticoids are the mainstay of the treatment. In clinical practice, the disease activity of PMR and corresponding treatment changes are based on the presence of symptoms and inflammatory markers. The interpretation of these abnormalities can be surprisingly difficult, especially when they are not consistent. In 2004, Leeb and Bird developed a composite score for measurement of disease activity in PMR, called the polymyalgia rheumatica activity score. It consists of 5 domains: morning stiffness time, ability to elevate the upper limbs, physician's global assessment, pain and CRP level. However, high-quality evidence on the measurement properties is lacking and there is still no consensus on the optimal cut off point.

Based on a Delphi study with physicians and patients OMERACT defines laboratory markers of systemic inflammation, pain, stiffness and physical function as the four inner core of domains considered mandatory for clinical trials of PMR, most frequently measured by erythrocyte sedimentation rate (ESR) and/or C-reactive protein (CRP), visual analogue scale (VAS) for pain, morning stiffness time and Health Assessment Questionnaire-Disability Index (HAQ-DI) respectively. Patient's global fatigue was strongly recommended to measure in PMR as well. Recently, a PMR-specific patient-reported outcome measure was developed, called the PMR impact scale. However, outcome measures in PMR studies lack consistency and there is no high-quality evidence on the measurement properties. In addition, the evolution of these patient reported outcomes is not known.

DETAILED DESCRIPTION:
The primary objective of this prospective observational trial is to validate the PMR-activity score and to determine the optimal cut-off point to discriminate between disease remission and active disease. The secondary objective is to assess the evolution of the patient reported outcomes during the disease course and their relation with disease activity.

The investigators intend to perform a 12-month, observational prospective trial in patients with recently diagnosed PMR. Patients will be followed and treated as standard of care. Follow-up visits will be planned at 8 weeks, 16 weeks, 26 weeks and 52 weeks. As in standard of care, additional visits can be planned if necessary, e.g. in case of symptoms suggestive of relapse. Each visit ESR, CRP, morning stiffness time, ability to elevate the upper limbs, physician's global assessment and VAS for pain as components of the PMR-activity score and VAS for global health, pain, stiffness and fatigue, HAQ-DI, Short Form Health survey (SF36) and PMR impact scale as patient-reported outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMR based on the judgment of an experienced clinician (affiliated with the general internal medicine or rheumatology department), taking into account all available information (clinical symptoms, biochemical, radiological, and PET results)
* Able to give informed consent
* Understanding and able to write Dutch, English or French

Exclusion Criteria:

* Concomitant diagnosis of giant cell arteritis (new diagnosis or being treated for giant cell arteritis)
* Concurrent rheumatoid arthritis, other inflammatory arthritis or other connective tissue disease
* Patients on glucocorticoids or other immunosuppressive drugs for another indication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of PMR
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Determination of the sensitivity and specificity of the PMR-activity score and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks

SECONDARY OUTCOMES:
Determination of the sensitivity and specificity of morning stiffness time and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of ability to elevate the upper limbs and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of physician's global assessment using a visual analogue scale and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of patient's assessment of pain using a visual analogue scale and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of C-reactive protein and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of the change in the PMR-activity score between two visits and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of the change in morning stiffness between two visits and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of the change in ability to elevate the upper limbs between two visits and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of the change in physician's global assessment using a visual analogue scale between two visits and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of the change in patient's assessment of pain using a visual analogue scale between two visits and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Determination of the sensitivity and specificity of the change in C-reactive protein between two visits and the optimal cut-off point to discriminate between disease remission and active disease | 52 weeks
Evolution of Health Assessment Questionnaire-Disability Index (HAQ-DI) over the disease course and the relation with disease activity | 52 weeks
Evolution of the ability to elevate the upper limbs over the disease course and the relation with disease activity | 52 weeks
Evolution of the patient's assessment of pain using a visual analogue scale over the disease course and the relation with disease activity | 52 weeks
Evolution of the patient's assessment of global health using a visual analogue scale over the disease course and the relation with disease activity | 52 weeks
Evolution of the patient's assessment of fatigue using a visual analogue scale over the disease course and the relation with disease activity | 52 weeks
Evolution of the patient's assessment of stiffness using a visual analogue scale over the disease course and the relation with disease activity | 52 weeks
Evolution of morning stiffness time over the disease course and the relation with disease activity | 52 weeks
Evolution of 36-item Short Form Health Survey (SF36) over the disease course and the relation with disease activity | 52 weeks
Evolution of the PMR impact scale over the disease course and the relation with disease activity | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vanderschueren, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leeb BF, Bird HA. A disease activity score for polymyalgia rheumatica. Ann Rheum Dis. 2004 Oct;63(10):1279-83. doi: 10.1136/ard.2003.011379. PMID 15361387
- [Background] Mackie SL, Twohig H, Neill LM, Harrison E, Shea B, Black RJ, Kermani TA, Merkel PA, Mallen CD, Buttgereit F, Mukhtyar C, Simon LS, Hill CL; OMERACT PMR Working Group. The OMERACT Core Domain Set for Outcome Measures for Clinical Trials in Polymyalgia Rheumatica. J Rheumatol. 2017 Oct;44(10):1515-1521. doi: 10.3899/jrheum.161109. Epub 2017 Aug 1. PMID 28765246
- [Background] Twohig H, Owen C, Muller S, Mallen CD, Mitchell C, Hider S, Hill C, Shea B, Mackie SL. Outcomes Measured in Polymyalgia Rheumatica and Measurement Properties of Instruments Considered for the OMERACT Core Outcome Set: A Systematic Review. J Rheumatol. 2021 Jun;48(6):883-893. doi: 10.3899/jrheum.200248. Epub 2020 Aug 1. PMID 32739892
- [Background] Twohig H, Mitchell C, Mallen CD, Muller S. Development and psychometric evaluation of the PMR-Impact Scale: a new patient reported outcome measure for polymyalgia rheumatica. Rheumatology (Oxford). 2023 Feb 1;62(2):758-765. doi: 10.1093/rheumatology/keac317. PMID 35639659